CLINICAL TRIAL: NCT00728650
Title: A Retrospective Review of Malignant Liver Tumors
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: TAB11119
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Liver Cancer
Keywords: hepatocellular carcinoma; colorectal carcinoma metastatic to liver; primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients with primary or metastatic hepatic malignancies

SUMMARY:
This study will review the treatment and outcomes of patients having primary and metastatic hepatic malignancies. Patients treated with surgical resection, percutaneous radiofrequency ablation (RFA), and transarterial chemoembolization (TACE) will be compared with patients not receiving these treatments. Tumor recurrence and survival data will be compared to the published literature to determine the efficacy of current treatment strategies in this patient population.

DETAILED DESCRIPTION:
Subjects will be identified by diagnosis and procedure codes from a university surgical practice and the St. John Medical Center Cancer Registry. Data will be obtained by review of both the clinic and hospital charts. In addition we plan to review and utilize liver tumor treatment and outcomes data from a national database. Treatment decisions, in cases managed by the primary investigator, were made on a clinical basis, often in collaboration with an interventional radiologist. Of the patients managed by the principal investigator, all procedures were undertaken after an informed consent process. Subjects were not exposed to risk beyond that posed by the recommended treatment. All treatments were within the scope of standard medical care. The primary investigator has no knowledge of the treatments chosen for the patients he did not manage. The subject's referring physician may be contacted to obtain follow-up data on the subject. The follow-up data will include: is the patient alive with disease; alive without disease, alive unknown; dead free of disease; dead with disease; dead unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or metastatic hepatic malignancies

Exclusion Criteria:

* Patients not diagnosed with primary or metastatic hepatic malignancies

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic and patients treated at St. John Medical Center in Tulsa, OK
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2003-10; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Survival | lifetime

SECONDARY OUTCOMES:
Efficacy | lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Broughan, MD, Principal Investigator — University of Oklahoma-Tulsa
Locations (1):
- The University of Oklahoma College of Medicine, Tulsa - Department of Surgery, Tulsa, Oklahoma, United States

REFERENCES:
- [Result] Curley SA, Izzo F, Delrio P, Ellis LM, Granchi J, Vallone P, Fiore F, Pignata S, Daniele B, Cremona F. Radiofrequency ablation of unresectable primary and metastatic hepatic malignancies: results in 123 patients. Ann Surg. 1999 Jul;230(1):1-8. doi: 10.1097/00000658-199907000-00001. PMID 10400029